CLINICAL TRIAL: NCT04687696
Title: Comparison of The Effects of Different Stretching Techniques in Overhead Athletes With Glenohumeral Internal Rotation Deficit
Brief Title: Comparison of The Effects of Different Stretching Techniques in Overhead Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gonca Şahiner Pıçak, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5003-GOA
Record Dates: First submitted 2020-12-22; First posted 2020-12-29 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Glenohumeral Internal Rotation Deficit

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post Isometric Relaxation Group (Experimental): The participants in this group will perform post isometric relaxation stretching in modified cross body position for 6 weeks.
  Interventions: Other: Post Isometric Relaxation Group
- Isolytic Stretching Group (Experimental): The participants in this group will perform isolytic stretching in modified cross body position for 6 weeks..
  Interventions: Other: Isolytic Stretching Group
- Static Stretching Group Group (Experimental): The participants in this group will receive static stretching in modified cross body position for 6 weeks.
  Interventions: Other: Static Stretching Group Group

INTERVENTIONS:
Other: Post Isometric Relaxation Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier barrier. The participants will be asked to perform an isometric contraction for 5 seconds in the horizontal abduction direction with 20% of the maximum muscle strength. After the relaxation, the arm will be moved towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between contractions.This stretching exercise will be applied in 5 repetitions in one session for 6 weeks 5 times a week.
  Arms: Post Isometric Relaxation Group
Other: Isolytic Stretching Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier barrier. The participants will be asked to perform a contraction in the horizontal abduction direction with 20% of the maximum muscle strength. When the muscle contraction occurs, the arm will be moved quickly in 2-4 seconds towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between stretches. This stretching exercise will be applied in 5 repetitions in one session for 6 weeks 5 times a week.
  Arms: Isolytic Stretching Group
Other: Static Stretching Group Group — Athletes will be positioned in a modified cross-body position. They will be asked to actively bring their underlying arm in the direction of horizontal adduction up to the physiological barrier. Then, the arm will be moved towards horizontal adduction and 15 seconds active-assistive stretching will be applied. Participants will be given a 5-second rest period between stretching exercises. This stretching exercise will be applied in 5 repetitions in one session for 6 weeks 5 times a week.
  Arms: Static Stretching Group Group

SUMMARY:
78 overhead athletes with Glenohumeral Internal Rotation Deficit (GIRD) will be included in this study. Participants will be randomly divided into 3 different groups of 26 people. In each group will be applied posterior shoulder stretching exercises (PSSE) performed with different Muscle Energy Techniques (MET).

DETAILED DESCRIPTION:
Post Isometric Relaxation Group (PIRG) participants will perform a PSSE with post isometric relaxation (PIR) technique, Isolytic Stretching Group (ISG) participants will perform a a PSSE with isolytic stretching technique and Static Stretching Group Group (SSG) participants will perform a PSSE with static stretching technique. All exercises will be performed in the modified crossbody position, for 5 times a week total of 6 weeks. Subacromial space, posterior capsule and muscle tendon thicknesses will be measured using a 7-12 MHz linear transducer with USG (LOGIQ e Ultrasound, GE Healthcare, USA). Athletes' GIRD results and rotational ROM measurements and Posterior shoulder tightness will be measured and recorded using a bubble inclinometer (Fabrication End Inc, New York, USA). Scapula kinematics (posterior tilt, upward rotation) will be evaluated with a digital inclinometer. Shoulder and scapular muscles will be evaluated with hend held dynamometer. Tightness of Levator scapulae and pectoralis minor will be assessed. The upper extremity functional performance of the athletes will be evaluated with the Functional Throwing Performance Index (FTPI). Evaluations will be performed before training program and repeated after 6 weeks of training, and at the 1st, 3th and 6th months after training program is completed and the effects of different muscle energy techniques (MET) will be compared. Investigators hypothesized 6 weeks of PSSE with different MET would have different effects on Acromio-Humeral Distance, posterior capsule thickness, muscle tendon thickness, rotational ROM measurements, scapula kinematics, muscle strength, posterior shoulder tightness and performance on overhead athletes with GIRD and the effects of MET would be superior to static stretching.

ELIGIBILITY:
Inclusion Criteria:

* Being overhead athlete
* Glenohumeral internal rotation range of motion of the affected shoulder should be less than other shoulder and bilateral shoulder internal rotation range of motion difference should be ≥15 º

Exclusion Criteria:

* Shoulder pain required medical attention for the last year.
* Current shoulder pain
* Cervical pain during upper extremity movement
* History of fracture to the shoulder girdle
* Systemic musculoskeletal disease
* History of shoulder surgery,
* Glenohumeral instability (positive apprehension, relocation, or positive sulcus test) or positive findings for a full thickness rotator cuff tear (positive lag sign, positive drop arm test, or marked weakness with shoulder external rotation)

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder internal rotation range of motion | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of shoulder internal rotation range of motion (with bubble inclinometer)

SECONDARY OUTCOMES:
Subacromial space | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of subacromial space ( with Ultrasound)
Posterior shoulder tightness | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of posterior shoulder tightness (with bubble inclinometer)
Shoulder Total rotation range of motion | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of shoulder internal rotation + external rotation range of motion (with bubble inclinometer)
Functional Throwing Performance Index | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Participants will throw a ball to shot a frame on a wall. Number of correct shots will be recorded.
Posterior capsule thickness | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of posterior capsule thickness ( with Ultrasound)
Muscle tendon thickness | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of supraspinatus, infraspinatus and teres minor tendon thicknesses ( with Ultrasound)
Scapula kinematics | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Posterior tilt and upward rotation of the scapula during arm elevation (with digital inclinometer)
Muscle Shortness | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Levator scapula and pectoralis minor shortness (with caliper and tape measure)
Eccentric strength | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of shoulder abduction and external rotation eccentric strength (in kg, with hand held dynamometer)
Isometric strength | baseline, 6 weeks of training, at the 1st, 3th and 6th months
  Change of lower trapezius muscle, serratus anterior and rotator cuff muscles isometric strength (in kg, with hand held dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi S Yeşilyaprak, Phd, Study Director — Dokuz Eylul University

IPD SHARING:
Plan to Share IPD: No